CLINICAL TRIAL: NCT00334867
Title: A Phase III Randomized Trial of Adding Vincristine-Topotecan-Cyclophosphamide to Standard Chemotherapy in Initial Treatment of Non-Metastatic Ewing Sarcoma
Brief Title: Combination Chemotherapy With or Without Topotecan in Treating Patients With Newly Diagnosed Localized Ewing's Sarcoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: withdrawn
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: AEWS0531; COG-AEWS0531 (Other: Children's Oncology Group); CDR0000483611 (Other: Clinical Trials.gov)
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Sarcoma
Keywords: localized Ewing sarcoma/peripheral primitive neuroectodermal tumor
MeSH Terms: conditions — Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Cyclophosphamide; Dexrazoxane; Doxorubicin; Etoposide; Ifosfamide; Topotecan; Vincristine; Radiotherapy

ARMS (2):
- Arm I (Active Comparator): Patients receive vincristine sulfate IV over 1 minute once a week on day 1 in weeks 1-3, 7-9, and 13-15; doxorubicin hydrochloride IV over 15 minutes on days 1 and 2 in weeks 1, 7, and 13; cyclophosphamide IV over 1 hour on day 1 in weeks 1, 7, and 13; and ifosfamide IV over 1 hour and etoposide IV over 1 hour on days 1-5 in weeks 4, 10, and 16. Patients undergo local therapy comprising conventional surgery (surgical resection) in approximately week 18 and/or radiation therapy beginning in approximately week 19.
  Interventions: Drug: cyclophosphamide; Drug: dexrazoxane hydrochloride; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: vincristine sulfate; Procedure: conventional surgery; Procedure: radiation therapy
- Arm II (Experimental): Patients receive vincristine sulfate IV over 1 minute once a week on day 1 in weeks 1-3, 7-9, and 13-16; topotecan hydrochloride IV over 30 minutes on days 1-5 in weeks 1 and 13; cyclophosphamide IV over 30 minutes on days 1-5 in weeks 1 and 13 and IV over 1 hour on day 1 in weeks 7 and 16; ifosfamide IV over 1 hour and etoposide IV over 1 hour on days 1-5 in weeks 4 and 10; and doxorubicin hydrochloride IV over 15 minutes on days 1 and 2 in weeks 7 and 16. Patients also undergo local therapy comprising of conventional surgery (surgical resection) in approximately week 18 and/or radiation therapy beginning in approximately week 19. Patients then proceed to combination chemotherapy.
  Interventions: Drug: cyclophosphamide; Drug: dexrazoxane hydrochloride; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: topotecan hydrochloride; Drug: vincristine sulfate; Procedure: conventional surgery; Procedure: radiation therapy

INTERVENTIONS:
Drug: cyclophosphamide — Given IV
Drug: dexrazoxane hydrochloride — Given IV
Drug: doxorubicin hydrochloride — Given IV
Drug: etoposide — Given IV
Drug: ifosfamide — Given IV
Drug: topotecan hydrochloride — Given IV
  Arms: Arm II
Drug: vincristine sulfate — Given IV
Procedure: conventional surgery — Patients undergo surgery in week 18
Procedure: radiation therapy — Patients undergo radiation therapy in week 19

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as vincristine, doxorubicin, cyclophosphamide, ifosfamide, etoposide, and topotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving chemotherapy after surgery may kill any tumor cells that remain after surgery. It is not yet known which combination chemotherapy regimen is more effective in treating Ewing's sarcoma.

PURPOSE: This randomized phase III trial is studying combination chemotherapy and topotecan to see how well they work compared with combination chemotherapy alone in treating patients with newly diagnosed localized Ewing's sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the event-free and overall survival of patients with newly diagnosed localized Ewing's sarcoma treated with doxorubicin hydrochloride, cyclophosphamide, vincristine, etoposide, and ifosfamide with vs without topotecan hydrochloride.
* Compare the side effects of these regimens in these patients.

Secondary

* Evaluate initial tumor size as a prognostic factor for event-free survival of these patients.
* Evaluate histological response as a prognostic factor for event-free survival of these patients.
* Continue evaluation of biologic markers both as related to prognosis and as eventual therapeutic targets via encouraging concurrent enrollment on COG-AEWS02B1.
* Evaluate radiologic response by positron emission tomography as a prognostic factor for event-free survival.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (≤ 17 vs ≥ 18 years of age) and primary tumor site (pelvic vs nonpelvic [including extra-osseous Ewing's sarcoma]). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive vincristine IV over 1 minute once a week on day 1 in weeks 1-3, 7-9, and 13-15; doxorubicin hydrochloride IV over 15 minutes on days 1 and 2 in weeks 1, 7, and 13; cyclophosphamide IV over 1 hour on day 1 in weeks 1, 7, and 13; and ifosfamide IV over 1 hour and etoposide IV over 1 hour on days 1-5 in weeks 4, 10, and 16. Patients undergo local therapy comprising surgical resection in approximately week 18 and/or radiotherapy beginning in approximately week 19. Patients then receive vincristine as above in weeks 19-21, 28-30, 34-36, 40-42, and 46-51; dexrazoxane hydrochloride IV over 15 minutes on days 1 and 2 and doxorubicin hydrochloride as above in weeks 19 and 28; cyclophosphamide as above in weeks 19, 28, 34, 40, 46, and 49; and ifosfamide and etoposide as above in weeks 22, 25, 31, 37, and 43.
* Arm II: Patients receive vincristine IV over 1 minute once a week on day 1 in weeks 1-3, 7-9, and 13-16; topotecan hydrochloride IV over 30 minutes on days 1-5 in weeks 1 and 13; cyclophosphamide IV over 30 minutes on days 1-5 in weeks 1 and 13 and IV over 1 hour on day 1 in weeks 7 and 16; ifosfamide IV over 1 hour and etoposide IV over 1 hour on days 1-5 in weeks 4 and 10; and doxorubicin hydrochloride IV over 15 minutes on days 1 and 2 in weeks 7 and 16. Patients undergo local therapy comprising surgical resection in approximately week 18 and/or radiotherapy beginning in approximately week 19. Patients then receive vincristine as above in weeks 19-21, 28-33, 37-42, and 46-48; topotecan hydrochloride as above in weeks 19, 31, and 40; cyclophosphamide IV over 30 minutes in weeks 19, 31, and 40 and IV over 1 hour in weeks 28, 37, and 46; ifosfamide and etoposide as above in weeks 22, 25, 34, 43, and 49; dexrazoxane hydrochloride IV over 15 minutes on days 1 and 2 in weeks 37 and 46; and doxorubicin hydrochloride as above in weeks 28, 37, and 46.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 528 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically and cytologically confirmed extracranial Ewing's sarcoma or primitive neuroectodermal tumor (PNET) of bone or soft tissue

  * Chest wall tumors with ipsilateral pleural effusions, ipsilateral positive pleural fluid cytology, or ipsilateral pleural-based secondary tumor nodules allowed

    * Contralateral pleural effusions or pleural nodules are not eligible
  * Tumor arising in the bony skull (extradural) are eligible

    * Tumors arising in the intradural soft tissue are not eligible
* Newly diagnosed disease

  * Only have had a biopsy of the primary tumor without an attempt at complete or partial resection
  * Prior attempted or accomplished unplanned excision allowed provided adequate imaging was obtained prior to surgery AND resection considered incomplete and further local control required
* No evidence of metastatic disease, defined as lesions discontinuous from the primary tumor, are not regional lymph nodes, and do not share a body cavity with the primary tumor
* No evidence of metastatic lung disease by CT scan

  * One pulmonary nodule > 1 cm in diameter OR > 1 nodule > 0.5 cm in diameter are considered evidence of pulmonary metastasis
  * Solitary nodules 0.5-1.0 cm or multiple nodules 0.3-0.5 cm must be confirmed negative by biopsy
  * Solitary nodules < 0.5 cm or multiple nodules < 0.3 cm not considered clear evidence of lung disease
* No distant nodule disease
* No esthesioneuroblastoma

PATIENT CHARACTERISTICS:

* Performance status (PS) 0-2 (Karnofsky PS 50-100% for patients ≥ 16 years of age or Lansky PS 50-100% for patients < 16 years of age)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥ 70 mL/min
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST or ALT < 2.5 times ULN
* Shortening fraction ≥ 27% by EKG
* Ejection fraction ≥ 50% by radionuclide angiogram
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiotherapy
* No prior chemotherapy

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2005-12; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Event-free survival

SECONDARY OUTCOMES:
Survival form study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Mason Bond, MD, Study Chair — Children's & Women's Hospital of British Columbia; Leo Mascarenhas, MD, Study Chair — Children's Hospital Los Angeles